CLINICAL TRIAL: NCT04219501
Title: Saving Time During Ventricular Arrhythmia Ablation With the Use of Non-Invasive ECG Imaging Technology
Brief Title: Ventricular Arrhythmia Ablation With the Use of Non-Invasive ECG Imaging Technology
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Mutual decision between the investigators and the sponsor
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Fred Kusumoto, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-007683
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Premature Ventricular Contraction; Ventricular Tachycardia
MeSH Terms: conditions — Ventricular Premature Complexes; Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Subjects presenting for PVC/VT ablation will undergo ablation procedures using standard of care invasive electroanatomical mapping systems.
- VIVO Arm (Experimental): Subjects presenting for PVC/VT ablation, that have a previously acquired cardiac CT/MRI scan or are having a cardiac CT/MRI scan as per routine care, will undergo ablation procedures using VIVO, a novel, non-invasive mapping system.
  Interventions: Other: VIVO

INTERVENTIONS:
Other: VIVO — Non-invasive mapping system software product that combines patient-specific images (MRI or CT) of the torso and cardiac structures and a 3D image of the torso that identifies precise ECG lead placement to generate a 3D model of the patient's heart.
  Arms: VIVO Arm

SUMMARY:
Researchers are trying to determine if the use of software called VIVO, made by Catheter Precision, Inc. can shorten the length of time it takes to perform an ablation procedure for either premature ventricular contractions (PVCs) and ventricular tachycardia (VT).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Structurally normal heart
* Cardiac MRI/CT as part of standard of care
* Diagnosed with premature ventricular contractions or ventricular tachycardia and scheduled to undergo an ablation to treat these conditions

Exclusion Criteria:

* Less than 18 years of age
* Structurally abnormal heart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Standard of care invasive electroanatomical mapping system duration | Baseline
  Total amount of time for standard of care invasive mapping measured in minutes
VIVO non-invasive mapping system duration | Baseline
  Total amount of time for non-invasive mapping using VIVO measured in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Fred Kusumoto, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials